CLINICAL TRIAL: NCT02961439
Title: Validation of Epworth Richmond's Echocardiography Education Focused Year
Acronym: VEREEFY
Status: Completed | Type: Observational
Sponsor: Epworth Healthcare (Other)
Collaborators: University of Melbourne (Other)
Responsible Party: Principal Investigator, Kyle Brooks, Intensivist, Epworth Healthcare
Other Study IDs: EH2016-133
Record Dates: First submitted 2016-11-03; First posted 2016-11-11 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Shock, Cardiogenic; Cardiac Tamponade; Pulmonary Embolism; Hypovolemia
MeSH Terms: conditions — Shock, Cardiogenic; Cardiac Tamponade; Pulmonary Embolism; Hypovolemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient Participants: Patient participants are adult patients in the Epworth Richmond Intensive care Unit. They are not the focus of the research but rather represent a general population of ICU patients that require echocardiography in the management of their critical illness. They will be a mix of medical and surgical patients some of whom are receiving mechanical ventilation, have movement restrictions, high BMI or other impediments to performing echocardiography.
- Registrar Participants: Registrar participants are doctors in training in ICU. They have completed a formal echo teaching program and completed a logbook of 30 supervised scans. They are the focus of the research and are being assessed on their diagnostic accuracy with echocardiography.
  Interventions: Behavioral: Epworth Richmond's Echocardiography Focused Year

INTERVENTIONS:
Behavioral: Epworth Richmond's Echocardiography Focused Year — a year long echo teaching program
  Groups: Registrar Participants

SUMMARY:
The use of echocardiography in intensive care is a developing field. In expert hands echocardiography has proven its utility in diagnosing cardiac pathology, differentiating shock states and in haemodynamic monitoring. However, whether the results obtained by experts can be generalized to trainees or specialists with limited training remains unclear. Further, concerns around training time and cost for intensive care staff have been a factor in limiting the uptake of echocardiography in intensive care.

The investigators aim to assess the diagnostic accuracy of Australian ICU doctors in training after completion of the current minimum training. After completing a structured teaching program and 30 mentored training scans trainees will be assessed on their accuracy with echocardiography. In the research phase trainees will complete a further 40 scans with each one matched with an expect scan. The results from the expert and trainee scans will be compared to determine the trainee's accuracy.

ELIGIBILITY:
Registrar Inclusion:

* At least 12 month appointment in Epworth Richmond ICU
* Completion of theoretical component of Epworth Richmond ICU echocardiography program
* Completion of 30 echocardiography scans

Registrar Exclusion:

• Previous experience in echocardiography prior to commencing at Epworth Richmond.

Patient Inclusion

* Patient in ICU or CCU
* 18 years or older
* Not likely to be discharged before completion of the scan

Patient Exclusion

* Likely to be discharged within next two hours
* Atrial fibrillation
* Presence of subcostal or intercostal drains or pneumothorax
* Unable to be consented
* Treating intensivist deems inclusion in study not suitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Registrar Participants and Patient Participant
Sampling Method: Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2016-11; Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Agreement between registrar and expert assessment of Left ventricular (LV) function | Four months

SECONDARY OUTCOMES:
Comparison of expert and registrar quantitative measures of Left vwentricular Internal Diameter in Diastole (LVIDd) | Four months
Comparison of expert and registrar quantitative measures of Left Ventricular Outflow Tract (LVOT) diameter | Four months
Comparison of expert and registrar quantitative measures of Left Ventricular Outflow Tract Velocity Time Integral (LVOT VTI) | Four months
Comparison of expert and registrar quantitative measures of TR V max | Four months
Comparison of expert and registrar quantitative measures of Tricuspid annular Plane Systolic Excursion (TAPSE) | Four months
Comparison of expert and registrar quantitative measures of IVC diameter | Four months
Comparison of expert and registrar qualitative assessment of pericardial fluid | Four months
Comparison of expert and registrar qualitative assessment of Left Ventricle : Right Ventricle size ratio | Four months

CONTACTS AND LOCATIONS:
Locations (1):
- Epworth Richmond, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Brooks KS, Tan LH, Rozen TH, Kelly D, McKenzie DP, Calafiore P, Barrett J. Validation of Epworth Richmond's Echocardiography Education Focused Year. Crit Care Med. 2020 Jan;48(1):e34-e39. doi: 10.1097/CCM.0000000000004076. PMID 31725442